CLINICAL TRIAL: NCT02726295
Title: The Efficacy of Mutaflor(E. Coli Nissle 1917, Mutaflor®) for Chronic Constipation:Multicenter Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-11-044-002
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E. coli Nissle 1917 (Mutaflor®) (Active Comparator): Mutaflor® group will receive E. coli Nissle 1917 (Mutaflor®) 28mg 2T tid for initial 2 days, then E. coli Nissle 1917, Mutaflor® 4T qd for the next 26 days.
  Interventions: Drug: E. coli Nissle 1917(Mutaflor®)
- Matched placebo (Placebo Comparator): Matched placebo group will receive placebo drug 28mg 2T tid for initial 2 days, then placebo 4T qd for the next 26 days. Placebo drug has same shape and size with E. coli Nissle 1917 (Mutaflor®).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E. coli Nissle 1917(Mutaflor®)
  Arms: E. coli Nissle 1917 (Mutaflor®)
Drug: Placebo
  Arms: Matched placebo

SUMMARY:
Chronic constipation is a prevalent, burdensome gastrointestinal disorder whose treatment remains challenging. There exist effective pharmacological therapies for chronic constipation, however, many patients do not well respond to current medications. Evidence suggests that disturbance in the gastrointestinal microbiota may be implicated in chronic constipation. Although, E.coli Nissle 1917 (Mutaflor®) has been used for chronic constipation, there are limited data regarding the efficacy of E.coli Nissle 1917 (Mutaflor®) in these patients. Therefore, this study aimed to investigate the efficacy of E.coli Nissle 1917 (Mutaflor®) in patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female outpatients aged from 20 to 75 years old.
* Patients meet International Congress of Gastroenterology (ROME III) clinical criteria for constipation*:

A. Must include two or more of the following:

1. Straining in > 1/4 defecations;
2. Lumpy or hard stools > 1/4 defecations;
3. Sensation of incomplete evacuation in 1/4 defecations;
4. Sensation of anorectal obstruction/blockage in > 1/4 defecations;
5. <3 defecations/week.

B.Loose stools are rarely present without the use of laxatives. C.There are insufficient criteria for irritable bowel syndrome. *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.

Exclusion Criteria:

* Pregnant or lactating woman
* Known organic gastrointestinal disease
* Subjects who diagnosed advanced adenoma within 3 years
* Prior gastrointestinal surgery (except appendectomy, herniotomy)
* Subjects who diagnosed irritable bowel syndrome
* Use of one or more of listed medications within 2 weeks (Laxative, Metoclopramide, Domperidone, Itopride, Levosulpride, Cisapride, Mosapride, Tegaserod, Prucalopride, Renzapride, Erythromycin, buspirone, Sumatriptan, Alosetron, Cilansetron, ondansetron, Citalopram, Paroxetine, Baclofen, Sildenafil, Nitroglycerin)
* Subjects who diagnosed lactulose malabsorption
* Subjects who diagnosed liver cirrhosis, severe congestive heart failure, severe renal insufficiency, uncontrolled hypertension, endocrine disorder, metabolic disorder, prior malignancy, immune deficiency
* Suspected obstruction, gastric retention, ileus, perforation, fecal impaction or inflammatory bowel disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Relief of constipation defined by improvement of complete spontaneous bowel movements(CSBMs/week) | 28days
  Subjects will report symptoms by questionnaire

SECONDARY OUTCOMES:
Improvement of average number of CSBMs/week | 28days
  Subjects will report symptoms by questionnaire
The time to 1st CSBM or SBM | 28days
  Subjects will report symptoms by questionnaire
Improvement of constipation related quality of life | 28days
  Subjects will report symptoms by questionnaire
Improvement of constipation related symptom | 28days
  Subjects will report symptoms by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Jin Lee, Professor, Principal Investigator — 56 Dalseong-Ro, Jung-Gu, Daegu, Korea; Jung Eun Shin, Professor, Study Director — Dankook Univ. Hospotal (31116) 201 Manghyang-ro, Dongnam-gu, Cheonan, Chung Nam, South Korea
Locations (1):
- Yoo Jin Lee, Daegu, South Korea